CLINICAL TRIAL: NCT00004063
Title: A Phase I-II Clinical Trial of Cisplatin (Platinol) Followed by Gemcitabine HCl (Gemzar) in Combination With Mild, Fever-Range Whole Body Hyperthermia (LL-WBH) at 40C in Patients With Advanced Malignancies
Brief Title: Cisplatin, Gemcitabine, Interferon Alfa, and Hyperthermia in Treating Patients With Advanced Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Joan M.C. Bull, University of Texas Health Science Center at Houston
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067264; UTHSC-MS-99116; NCI-V99-1561; NCT00005929 (obsolete NCT alias)
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2008-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Interferon-alpha; Cisplatin; Gemcitabine; Diathermy

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: cisplatin
Drug: gemcitabine hydrochloride
Procedure: hyperthermia treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of cancer cells. Hyperthermia therapy kills tumor cells by heating them to several degrees above body temperature. Combining hyperthermia with chemotherapy and interferon alfa may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects of cisplatin, gemcitabine, interferon alfa, and whole-body hyperthermia and how well they work in treating patients with metastatic, recurrent, or refractory cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity and tumor response in patients with metastatic, recurrent, or refractory malignancies treated with cisplatin, gemcitabine, interferon alfa, and long-duration, low temperature whole body hyperthermia (LL-WBH).

OUTLINE: This is a dose escalation study of cisplatin.

* Phase I and II: Patients receive gemcitabine IV over 30 minutes on day 1 and 8. Patients receive cisplatin IV over 6 hours on day 15, followed by subcutaneous interferon alfa on days 16 and 17. Patients undergo long-duration, low temperature whole body hyperthermia over 6 hours plus gemcitabine over 30 minutes on day 17. Courses repeat every 5 weeks in the absence of disease progression or unacceptable toxicity.
* Phase I: Cohorts of 3-6 patients receive escalating doses of cisplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose limiting toxicity. The MTD of cisplatin is used for phase II study.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic, recurrent, or refractory carcinoma
* Measurable disease by CT, MRI, or physical examination
* No brain metastases or other CNS disorders

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 90,000/mm^3
* Bone marrow cellularity normal on bone marrow biopsy
* No coagulopathy disorder

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT no greater than 2 times upper limit of normal
* PT less than 14 seconds
* PTT less than 35 seconds
* No inadequate liver function (no greater than 20% involvement)

Renal:

* Creatinine no greater than 1.8 mg/dL
* Creatinine clearance at least 45 mL/min
* BUN no greater than 25 mg/dL

Cardiovascular:

* Adequate cardiac function documented by history, physical exam, or stress exercise test (MUGA or ECHO) with resting blood pressure and heart rate increasing appropriately with exercise
* LVEF at least 45%
* No prior myocardial infarction
* No symptomatic coronary artery disease
* No angina
* No significant arrhythmia
* No uncontrolled hypertension
* No thromboembolic disease

Pulmonary:

* FEV_1 at least 70% of predicted
* Arterial PO_2 at least 60 mmHg on room air
* No massive (greater than 30% involvement) lung disease
* DLCO greater than 50% of predicted

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No seizure disorders
* No significant emotional instability
* No history of malignant hyperthermia following general anesthesia
* No other concurrent medical illness that would prevent compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* At least 6 days since major thoracic or abdominal surgery

Other:

* No concurrent cardiac glycosides, antiangina drugs, arrhythmia drugs, anticoagulants, thrombolytic agents, adrenal corticosteroids, or aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1999-08; Primary Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Response duration
Duration of stable disease
Overall survival
Progression-free survival
Time to response

CONTACTS AND LOCATIONS:
Overall Officials: Joan M.C. Bull, MD, Study Chair — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States